CLINICAL TRIAL: NCT00953784
Title: Minimization of Surgical Site Infections for Pts Undergoing Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Thomas Anthony, MD Chief of Surgery, VANTXHCS Dallas, TX
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-025
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-05

CONDITIONS: Surgical Wound Infections; Colorectal Surgery
Keywords: surgery; wound infections; colorectal
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard management
- 2 (Active Comparator): Extended management: with no bowel prep except enema,restricted fluids, increased O2,body warming and use of skin protectors during surgery as previously described
  Interventions: Procedure: standard operating management

INTERVENTIONS:
Procedure: standard operating management — As previously described
  Other Names: Extended management
  Arms: 2

SUMMARY:
This is a comparison, at this VA Hospital, of standard operating room management in colorectal surgery to a more rigid management using an additional five previously tested treatments to determine if this changes the rate of post operative wound infections.

DETAILED DESCRIPTION:
A comparison between standard operating room:

1. use of pre-op bowel prep (Golytely or Phosphosoda,plus 3 doses of oral antibiotics(Erythromycin and Neomycin), and fleets enema the day before surgery
2. Standard anesthesia FiO2 (approx. 30-50%)during surgery
3. Standard IV fluids during surgery(greater than 200cc per hour)
4. Standard post-op O2 by mask for 2 hours

To extended operating room procedures of:

1. No po antibiotics or pre-op bowel prep other than enema prior to surgery
2. Skin warming at least 15 minutes prior to and during surgery(core temp 36C+)
3. IOBAN drapes and Plastic wound protectors used during surgery
4. Restricted IV fluids less than 200cc per hour during surgery
5. Increased FiO2 to 80% during surgery and 2 hours after by mask

Monitoring for post-op wound infections at discharge and up to 30days post-op

ELIGIBILITY:
Inclusion Criteria:

* Scheduled VA adult elective colorectal surgery patient

Exclusion Criteria:

* Non VA adults, emergent colorectal surgery, scheduled multiple surgery procedures,pts with other infections being treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
%/type Surgical wound infections rated per infection classifications of NNIS/CDC | with in 30 days post-op

SECONDARY OUTCOMES:
%/type surgical wound infections per classifications per NNIS/CDC | at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: James LePage, Ph.D, Study Chair — ACOS for Research VANorth Tx Health Care System
Locations (1):
- VA North Texas Health Care System, Dallas, Texas, United States

REFERENCES:
- [Derived] Anthony T, Murray BW, Sum-Ping JT, Lenkovsky F, Vornik VD, Parker BJ, McFarlin JE, Hartless K, Huerta S. Evaluating an evidence-based bundle for preventing surgical site infection: a randomized trial. Arch Surg. 2011 Mar;146(3):263-9. doi: 10.1001/archsurg.2010.249. Epub 2010 Nov 15. PMID 21079110
- See also: homepage — http://www.northtexas.va.gov/